CLINICAL TRIAL: NCT02072304
Title: Study of Web-based Cognitive Behavioral Therapy in Adolescent Depression; Randomized Controlled Trial for Korean Adolescents
Brief Title: Study of Web- Based Cognitive Behavioral Therapy for Depressed Korean Adolescents
Acronym: wogyeokdajim
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Ju Hong, associate professor department of psychiatry, Hallym University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-001
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Depression; Mental Disorder in Adolescence; Cognitive Behavioral Therapy
Keywords: mood disorder; depressive disorder; mental disorders; program acceptability; behavioral symptoms; suicidal ideation; patient adherence
MeSH Terms: conditions — Depression; Mood Disorders; Depressive Disorder; Mental Disorders; Behavioral Symptoms; Suicidal Ideation; Patient Compliance | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- web-based CBT (Experimental): Web-based CBT group : The intervention is made up of 8 internet modules based on behavioral activation, cognitive behavioral therapy
  Interventions: Behavioral: web-based CBT
- supportive care (Active Comparator): supportive care group will receive supportive care for treating depression by e-mail per a week for 8 weeks
  Interventions: Behavioral: supportive care

INTERVENTIONS:
Behavioral: web-based CBT — A cognitive behavioral program in 8 weeks that will provide participants with the following: online interactive tools to do their homeworks and guidance on using cognitive and behavioral strategies to help reduce depressive symptoms, information about the depressive symptoms and cognitive behavioral therapy
  Other Names: wogyeokdajim
  Arms: web-based CBT
Behavioral: supportive care — supportive care group will receive supportive care for treating depression by e-mail per a week for 8 weeks with the following: psychoeducation about depression, stigma of mental illness, distraction technique, emotional regulation, active scheduling.
  Other Names: supportive care for depressed adolescents
  Arms: supportive care

SUMMARY:
The purpose of this study is to develope web-based cognitive behavioral therapy for Korean adoldescents who have a mild depression. And we will investigate whether web-based cognitive behavioral therapy is more effective than supportive psychotherapy for treating depressed adolescents. Our hypothesis is web- based cognitive behavioral is more effective than supportive psychotherapy

DETAILED DESCRIPTION:
We will recruit adolescents(age 12-18 years old) with a diagnosis of major depressive disorder, dysthymia and depressive disorder NOS in outpatient clinic of child and adolescent psychiatry and we will advertise for recruitment of subjects in community. The study protocol will be approved by the Institutional Review Board of the Hallym university sacred heart hospital. Well- trained interviewers will conduct the assessments of participants and their parents or guardians. The assessment included the diagnostic interview, demographic characteristics, depressive symptom severity scale , Columbia suicide severity rating scale, questionnaire about abuse histories.

We decided the number of participants of 164, because in previous studies, web- based cognitive behavioral therapy showed mild to moderate effect size (effect size = 0.43). So for examining the hypothesis, we will recruit 164 adolescents by calculating the number of participants using G power program version 3.1.3. (level of significance = 5%, power of a hypothesis test = 80%, drop out rate = 20%)

And we will conduct randomized controlled trial for examining the efficacy of web- based cognitive behavioral therapy. Our hypothesis is web- based cognitive behavioral is more effective than supportive psychotherapy, so we will deliver web- based cognitive behavioral therapy program to cognitive behavioral therapy group for 8 weeks(once in a week), and supportive psychotherapy to supportive psychotherapy group for 8 weeks(once in a week) We will exclude the participant if the participant has severe depressive symptoms, definite suicidal idea, plan and attempt, psychotic symptoms, bipolar disorders, sexual abuse histories, other neurological diseases or received cognitive behavioral therapy, pharmacotherapy or interpersonal psychotherapy.

We will analyze the intent- to- treat population. For each individual, missing values are replaced by the last observed value of that variable. And we will use Chi square test or repeated measure-ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of major depressive disorder, dysthymic disorder and depressive disorder NOS
* participants and their parents both agree informed consents

Exclusion Criteria:

* participants have psychotic symptoms, developmental disorders,
* participants are diagnosed by bipolar disorder
* participants are current high risk of suicide
* participants have psychiatric and physical symptoms need urgent medicine treatment
* participants have a history of sexual abuse
* participants have cognitive behavioral therapy or interpersonal psychotherapy within 3 months
* participants have a history of brain injury or a neurological disorder such as seizure disorder, or severe physical disorder

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 164 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
The Center for Epidemiological Studies of Depression (CES-D) Scale | 0, 4, 8 weeks
  Change in CESD from baseline Change in CESD scale between and within groups across the 8 weeks and for each assessment point
Subjective depressed mood scale | each week during 8 weeks
  Change in Subjective depressed mood scale from baseline Change in Subjective depressed mood scale scale within web CBT groups across the 8 week
The Korean youth self report (K-YSR) | 0, 8 weeks
  Change in K-YSR from baseline Change in K-YSR scale between and within groups across the 8 weeks

SECONDARY OUTCOMES:
Acceptability and adherence of Web-based cognitive behavioral treatment program for adolescents with depression | 8 weeks
  After treatment, we will check out how many the participants complete the session.
satisfaction of Web-based cognitive behavioral treatment program of both adolescents with depression and their parents | 8 week
  After treatment, we will check out how the participants and their parent feel satisfaction about treatment
Columbia suicide severity rating scale | 0, 4 8 weeks after baseline assessment
  Change in CSSRS from baseline Change in CSSRS scale between and within groups across the 8 weeks and for each assessment point
Adolescent's characteristics that moderate the impact of the program | 0, 4 and 8 weeks after baseline assessment
  we will find out adolescent's characteristics that moderate the impact of the program

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-ju hong, MD PHD, Principal Investigator — Associate Professor of Department of Psychiatry of Hallym University Sacred Heart Hospital
Locations (3):
- South Korea (3):
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - National health insurance service ilsan hospital, Goyang-si, Gyeonggi-do
  - Inje university ilsan paik hospital, Goyang-si, Gyeonggi-do

REFERENCES:
- [Background] Angold A, Messer SC, Stangl D, Farmer EM, Costello EJ, Burns BJ. Perceived parental burden and service use for child and adolescent psychiatric disorders. Am J Public Health. 1998 Jan;88(1):75-80. doi: 10.2105/ajph.88.1.75. PMID 9584037
- [Background] Brent DA, Perper JA, Goldstein CE, Kolko DJ, Allan MJ, Allman CJ, Zelenak JP. Risk factors for adolescent suicide. A comparison of adolescent suicide victims with suicidal inpatients. Arch Gen Psychiatry. 1988 Jun;45(6):581-8. doi: 10.1001/archpsyc.1988.01800300079011. PMID 3377645
- [Background] Birmaher B, Ryan ND, Williamson DE, Brent DA, Kaufman J, Dahl RE, Perel J, Nelson B. Childhood and adolescent depression: a review of the past 10 years. Part I. J Am Acad Child Adolesc Psychiatry. 1996 Nov;35(11):1427-39. doi: 10.1097/00004583-199611000-00011. PMID 8936909
- [Background] Bostwick JM, Pankratz VS. Affective disorders and suicide risk: a reexamination. Am J Psychiatry. 2000 Dec;157(12):1925-32. doi: 10.1176/appi.ajp.157.12.1925. PMID 11097952
- [Background] Birmaher B, Brent D; AACAP Work Group on Quality Issues; Bernet W, Bukstein O, Walter H, Benson RS, Chrisman A, Farchione T, Greenhill L, Hamilton J, Keable H, Kinlan J, Schoettle U, Stock S, Ptakowski KK, Medicus J. Practice parameter for the assessment and treatment of children and adolescents with depressive disorders. J Am Acad Child Adolesc Psychiatry. 2007 Nov;46(11):1503-26. doi: 10.1097/chi.0b013e318145ae1c. PMID 18049300
- [Background] March J, Silva S, Petrycki S, Curry J, Wells K, Fairbank J, Burns B, Domino M, McNulty S, Vitiello B, Severe J; Treatment for Adolescents With Depression Study (TADS) Team. Fluoxetine, cognitive-behavioral therapy, and their combination for adolescents with depression: Treatment for Adolescents With Depression Study (TADS) randomized controlled trial. JAMA. 2004 Aug 18;292(7):807-20. doi: 10.1001/jama.292.7.807. PMID 15315995
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] Van Voorhees BW, Vanderplough-Booth K, Fogel J, Gladstone T, Bell C, Stuart S, Gollan J, Bradford N, Domanico R, Fagan B, Ross R, Larson J, Watson N, Paunesku D, Melkonian S, Kuwabara S, Holper T, Shank N, Saner D, Butler A, Chandler A, Louie T, Weinstein C, Collins S, Baldwin M, Wassel A, Reinecke MA. Integrative internet-based depression prevention for adolescents: a randomized clinical trial in primary care for vulnerability and protective factors. J Can Acad Child Adolesc Psychiatry. 2008 Nov;17(4):184-96. PMID 19018321
- [Background] Van Voorhees BW, Fogel J, Reinecke MA, Gladstone T, Stuart S, Gollan J, Bradford N, Domanico R, Fagan B, Ross R, Larson J, Watson N, Paunesku D, Melkonian S, Kuwabara S, Holper T, Shank N, Saner D, Butler A, Chandler A, Louie T, Weinstein C, Collins S, Baldwin M, Wassel A, Vanderplough-Booth K, Humensky J, Bell C. Randomized clinical trial of an Internet-based depression prevention program for adolescents (Project CATCH-IT) in primary care: 12-week outcomes. J Dev Behav Pediatr. 2009 Feb;30(1):23-37. doi: 10.1097/DBP.0b013e3181966c2a. PMID 19194326
- [Background] Calear AL, Christensen H, Mackinnon A, Griffiths KM, O'Kearney R. The YouthMood Project: a cluster randomized controlled trial of an online cognitive behavioral program with adolescents. J Consult Clin Psychol. 2009 Dec;77(6):1021-32. doi: 10.1037/a0017391. PMID 19968379
- [Background] Posner K, Oquendo MA, Gould M, Stanley B, Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. Am J Psychiatry. 2007 Jul;164(7):1035-43. doi: 10.1176/ajp.2007.164.7.1035. PMID 17606655